CLINICAL TRIAL: NCT04701463
Title: Effect of a Specialized Amino Acid Mixture on Body Composition and Skin State in Overweight and Obese Class I Sedentary Postmenopausal Women
Brief Title: A Specialized Amino Acid Mixture on Body Composition and Skin State in Overweight and Obese Class I Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0912/14122018
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Amino Acid; Body Weight Changes; Skin Manifestations; Obesity; Postmenopausal Disorder
MeSH Terms: conditions — Body Weight Changes; Skin Manifestations; Obesity | interventions — Glutamine; Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-glutamine, L-arginine and calcium beta-hydroxy-beta-methylbutyrate supplement (Experimental)
  Interventions: Dietary Supplement: L-glutamine, L-arginine and calcium beta-hydroxy-beta-methylbutyrate
- Placebo (Placebo Comparator)
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Dietary Supplement: L-glutamine, L-arginine and calcium beta-hydroxy-beta-methylbutyrate — 2 daily sachets (mid morning and mid afternoon) of an oral dietary supplement with L-glutamine and L-arginine and calcium beta-hydroxy-beta-methylbutyrate
  Arms: L-glutamine, L-arginine and calcium beta-hydroxy-beta-methylbutyrate supplement
Combination Product: Placebo — Isocaloric formula
  Arms: Placebo

SUMMARY:
The use of dietary amino acids has been explored for therapeutic and safety intervention of obesity and obesity-induced dysfunction. In particular, 3 molecules have been shown to be effective both in the animal model and in humans, in promoting the loss of fat mass, specifically visceral adipose tissue, and in maintaining free fat mass: arginine, glutamine and leucine (and its metabolite beta hydroxy methyl butyrate, HMB). The aim of this study was to evaluate the efficacy in terms of fat mass, in particular Visceral Adipose Tissue reduction, as primary end point, in obese patients following the administration of specific food for special medical purposes (FSMP) for muscle recovery, consisting of arginine, glutamine and HMB. The secondary end point is the evaluation of skin state, by a validate self-reported questionnaire survey to assess skin, after 4- weeks intake of this FSMP.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopause
* Obesity (I class) or overweight

Exclusion Criteria:

* Taking any medication
* Having liver, renal and thyroid disease
* Smoking
* Drinking more than two standard alcoholic beverages/day (20 g of alcohol/day)

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Changes on Visceral Adipose Tissue | Baseline / 30 days
  Evaluation of Visceral Adipose Tissue (g)

SECONDARY OUTCOMES:
Changes on Body Composition | Baseline / 30 days
  Evaluation of fat mass and fat free mass (g)
Changes on Metabolic parameters | Baseline / 30 days
  Evaluation of Fasting blood glucose (mg/dl), total cholesterol (mg/dl), low-density lipoprotein-cholesterol (mg/dl), high-density lipoprotein-cholesterol (mg/dl) and triglyceride levels (mg/dl)
Changes on Metabolic parameters | Baseline / 30 days
  Evaluation of insulin (mcIU/mL)
Changes on Metabolic parameters | Baseline / 30 days
  Evaluation of insulin resistance (HOMA index)
Changes on anthropometric measurements | Baseline / 30 days
  Evaluation of body weight (kg) and height (m) combined for Body Mass Index (kg/m2)
Changes on anthropometric measurements | Baseline / 30 days
  Evaluation of waist circumference (cm)
Changes on skin condition | Baseline / 30 days
  Administration of a questionnaire survey with a point evaluation scale from 0 to 5 (Oe et al, 2017). For the skin luster and suppleness, one is the worst and five is the best. For the wrinkles, one is least wrinkles; not worry, and five is most wrinkles; most care.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda di Servizi alla Persona, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No